CLINICAL TRIAL: NCT01202916
Title: Quality of Life Among Children With Congenital Heart Disease
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: 8422
Record Dates: First submitted 2010-09-14; First posted 2010-09-16 (Estimated); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Congenital Heart Disease
Keywords: children with congenital heart disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Congenital Heart Disease
- Healthy children

SUMMARY:
Congenital heart diseases (CHD) are the first cause of congenital malformations with an incidence of 8 for 1000 births. Within the two past decades prenatal diagnosis has had a great impact on CHD prevalence. France was the first country to show the impact of prenatal diagnosis on the lowering prevalence of the most severe CHD, the hypoplastic left heart syndrome. Since the 90's, great advances in pediatric cardiac surgery, intensive care and cardiac catheterization have led to lower mortality and morbidity in this population. Prevalence of " GUCH ", grown-ups with congenital heart disease has thus been significantly increasing. For all these reasons and as the investigators can also see in other many chronic diseases, new questions about the quality of life of these patients arise among patients, parents/future parents, doctors, patients associations, and public health organizations. In 2007 French government promoted a national public health plan for "improvement of the quality of life among patients suffering from chronic illnesses". First step of such a program is to correctly evaluate this quality of life. Indeed the concept of "quality of life" (QoL) remains subjective and difficult to appreciate and measure. Its analysis requires the use of validated questionnaires. Few questionnaires are available in Europe, especially in pediatrics. Few studies in this population have been led and no comparative study to a control randomized group has been published. The investigators study aims to analyze in the investigators tertiary care center in pediatric cardiology the QoL among 8 to 18 year old French patients with CHD using a validated questionnaire (Kidscreen™) and to compare it to same aged healthy children. The investigators secondarily intend to :- validate the French version of one reference pediatric QoL questionnaire used in most publications in the USA (PedsQL™). - compare the QoL to the severity of the CHD using a published semi-quantitative score.- compare the QoL to the severity of the CHD using the results of routine exercise tests (VO2 max) performed routinely in the investigators center. The investigators hypothesis are that :- Quality of life of most common and not severe CHD is close to that of healthy children. - QoL of severe CHD is not so well correlated to severity of CHD.- PedsQL™ is a simple questionnaire which can be used in France in routine follow-up of children with CHD.

ELIGIBILITY:
Inclusion Criteria:

* patients with congenital heart disease (defined by Chapter Q of the ICD-10)
* Patient participation in the study noted in the medical record.Exclusion Criteria:
* Age greater than or equal to 8 years and less than 18 years
* Whose parents signed written consent
* Obligation of membership or beneficiary of a French social security

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: * children with congenital heart disease
  * healthy children
Sampling Method: Non-Probability Sample
Enrollment: 316 (Actual)
Dates: Start 2009-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Quality of Life questionnaire | one day

CONTACTS AND LOCATIONS:
Overall Officials: AMEDRO Pascal, MD, PhD, Principal Investigator — UH Montpellier
Locations (1):
- Pediatric and Congenital Cardiology and Pulmonology Department, Arnaud De Villeneuve University Hospital, Montpellier, France

REFERENCES:
- [Background] Amedro P, Tahhan N, Bertet H, Jeandel C, Guillaumont S, Mura T, Picot MC. Health-related quality of life among children with Turner syndrome: controlled cross-sectional study. J Pediatr Endocrinol Metab. 2017 Aug 28;30(8):863-868. doi: 10.1515/jpem-2017-0026. PMID 28753541
- [Background] Amedro P, Bajolle F, Bertet H, Cheurfi R, Lasne D, Nogue E, Auquier P, Picot MC, Bonnet D. Quality of life in children participating in a non-selective INR self-monitoring VKA-education programme. Arch Cardiovasc Dis. 2018 Mar;111(3):180-188. doi: 10.1016/j.acvd.2017.05.013. Epub 2017 Nov 1. PMID 29100908
- [Result] Amedro P, Dorka R, Moniotte S, Guillaumont S, Fraisse A, Kreitmann B, Borm B, Bertet H, Barrea C, Ovaert C, Sluysmans T, De La Villeon G, Vincenti M, Voisin M, Auquier P, Picot MC. Quality of Life of Children with Congenital Heart Diseases: A Multicenter Controlled Cross-Sectional Study. Pediatr Cardiol. 2015 Dec;36(8):1588-601. doi: 10.1007/s00246-015-1201-x. Epub 2015 May 31. PMID 26024647
- [Result] Gavotto A, Vandenberghe D, Abassi H, Huguet H, Macioce V, Picot MC, Guillaumont S, Matecki S, Amedro P. Oxygen uptake efficiency slope: a reliable surrogate parameter for exercise capacity in healthy and cardiac children? Arch Dis Child. 2020 Dec;105(12):1167-1174. doi: 10.1136/archdischild-2019-317724. Epub 2020 Jul 30. PMID 32732318
- [Result] Amedro P, Gavotto A, Guillaumont S, Bertet H, Vincenti M, De La Villeon G, Bredy C, Acar P, Ovaert C, Picot MC, Matecki S. Cardiopulmonary fitness in children with congenital heart diseases versus healthy children. Heart. 2018 Jun;104(12):1026-1036. doi: 10.1136/heartjnl-2017-312339. Epub 2017 Nov 23. PMID 29170358
- [Result] Abassi H, Gavotto A, Picot MC, Bertet H, Matecki S, Guillaumont S, Moniotte S, Auquier P, Moreau J, Amedro P. Impaired pulmonary function and its association with clinical outcomes, exercise capacity and quality of life in children with congenital heart disease. Int J Cardiol. 2019 Jun 15;285:86-92. doi: 10.1016/j.ijcard.2019.02.069. Epub 2019 Mar 1. PMID 30857849
- [Result] Gavotto A, Huguet H, Picot MC, Guillaumont S, Matecki S, Amedro P. The V̇e/V̇co2 slope: a useful tool to evaluate the physiological status of children with congenital heart disease. J Appl Physiol (1985). 2020 Nov 1;129(5):1102-1110. doi: 10.1152/japplphysiol.00520.2020. Epub 2020 Sep 10. PMID 32909919
- [Result] Amedro P, Huguet H, Macioce V, Dorka R, Auer A, Guillaumont S, Auquier P, Abassi H, Picot MC. Psychometric validation of the French self and proxy versions of the PedsQL 4.0 generic health-related quality of life questionnaire for 8-12 year-old children. Health Qual Life Outcomes. 2021 Mar 4;19(1):75. doi: 10.1186/s12955-021-01714-y. PMID 33663527
- [Derived] Amedro P, Picot MC, Moniotte S, Dorka R, Bertet H, Guillaumont S, Barrea C, Vincenti M, De La Villeon G, Bredy C, Soulatges C, Voisin M, Matecki S, Auquier P. Correlation between cardio-pulmonary exercise test variables and health-related quality of life among children with congenital heart diseases. Int J Cardiol. 2016 Jan 15;203:1052-60. doi: 10.1016/j.ijcard.2015.11.028. Epub 2015 Nov 10. PMID 26638054